CLINICAL TRIAL: NCT05623176
Title: Improvement in Patient Survival and Equality in Care Provision for General Surgery Patients Undergoing Emergency Laparotomy - Can This be Achieved Through the Implementation of Standardised Care Protocols?
Brief Title: Clinical Outcomes and Equality in Healthcare for Emergency General Surgery Patients Undergoing Emergency Laparotomy
Acronym: LAPTOP
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Rebecka Ahl Hulme, Principal investigator, Region Stockholm
Other Study IDs: K2022-9097
Record Dates: First submitted 2022-11-12; First posted 2022-11-21 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Abdomen, Acute
Keywords: Emergency laparotomy; General surgery; Clinical outcomes
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Old routine of non-standardised laparotomy care: Group following the old routine of emergency laparotomy care i.e. no existing standardised care protocols.
- New routine of standardised laparotomy care: Group which has been part of the hospital's new standardised care routine for emergency laparotomy.
  Interventions: Other: Standardised laparotomy care

INTERVENTIONS:
Other: Standardised laparotomy care — This is a cohort study and no intervention as part of the study has been introduced. We are studying two groups and comparing the two before and after the introduction of a standardised laparotomy care protocol as part of a clinical quality improvement measure.
  Groups: New routine of standardised laparotomy care

SUMMARY:
The goal of this observational cohort study is to evaluate the standard of care for general surgerical patients undergoing emergency laparotomy and assess factors affecting clinical outcomes, as well as evaluating the quality of life in the year after abdominal surgery.

The main questions it aims to answer are:

1. what factors are associated with adverse post-operative events
2. are patients treated differently based on sex or age
3. how does quality of life look like and possibly change over the coarse of a year after surgery

This is an evaluation of the current standard of care and the outcomes of this patient group prior to the implementation of a standardised care protocols for emergency laparotomy patients. Secondly, the study aims to, over time, compare results before and after the introduction of this standardised care protocol.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing emergency laparotomy due to general surgical indication

Exclusion Criteria:

* Children under 16
* Trauma laparotomy
* Vascular, urological or gynaecological indication for laparotomy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion of adult general surgical patients undergoing an emergency laparotomy during period 2015 and 2029. The cohort of 2015-2022 will be compared to the cohort of 2023-2029 in terms of general outcomes. The cohort of 2023-2029 will specifically be studied for any impact of emergency laparotomy on quality of life.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 30 days

SECONDARY OUTCOMES:
In-hospital serious complications | 30 days
  Severity measured through Clavien-Dindo classification
Long-term mortality | 1 year
Quality of life questionnaires | 1 year
  As measured through questionnaires at 1 month, 3 months and up to 1 year post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecka Ahl Hulme, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden